CLINICAL TRIAL: NCT04893980
Title: Short-term Efficacy of Low-dose Interleukin-2 Treatment in Chrornic Spontaneous Urticaria: a Randomized, Controlled, Single-center Clinical Trial
Brief Title: Efficacy of Low-dose Interleukin-2 Treatment in Chronic Spontaneous Urticaria
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Qianjin Lu, MD, PhD, Professor and Director, Institute of Dermatology, Central South University, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSU202009
Record Dates: First submitted 2021-01-31; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: chronic urticaria; interleukin-2
MeSH Terms: conditions — Chronic Urticaria | interventions — aldesleukin; Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-dose interleukin-2 treatment group (Experimental): Use Interleukin-2 to treat CSU during day1-day28.
  Interventions: Drug: Recombinant human interleukin-2 (rhIL-2)
- Control group (Other): Use Interleukin-2 to treat CSU during day15-day28.
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: Recombinant human interleukin-2 (rhIL-2) — During Day 0-14, patients in this group will receive treatment with antihistamines at the same dosage as pre-recruitment, together with a low-dose recombinant human Interleukin-2 (rhIL-2) at a dosage of 1 million international units every other day by intramuscular injection (rhIL-2, 1 MIU, im, Qod). During Day 15-28, the injections of rhIL-2 will be continued at the same dosage and the dose of antihistamines may be adjusted according to the control of symptoms.
  Other Names: Recombinant Human Interleukin-2 (I)
  Arms: Low-dose interleukin-2 treatment group
Drug: Control group — During Day 0-14, patients in the control group receive treatment with only antihistamines at the same dosage as pre-recruitment, but no injection of rhIL-2. During Day 15-28, treatment with low dose recombinant human Interleukin-2 (rhIL-2), i.e., 1 million international units every other day by subcutaneous or intramuscular injection (rhIL-2, 1MIU, im, Qod), will be added.
  Other Names: No injections during Day 0-14
  Arms: Control group

SUMMARY:
This study is a randomized, controlled, single-center clinical study to evaluate the short-term efficacy of low-dose Interleukin-2 injection as an add-on therapy for the treatment of patients aged 18-75 who have been diagnosed with CSU and remain symptomatic despite oral antihistamine treatment .

DETAILED DESCRIPTION:
Backgrounds:

Urticaria is a common disorder that present with localized edema reaction caused by dilatation and increased permeability of small blood vessels in skin and mucosa. The main clinical manifestations are wheal and erythema reaction.

Chronic spontaneous urticaria (CSU) is defined as the recurrent, transient (<24h), pruritic wheals of the skin and mucosa lasting for more than 6 weeks ,with or without angioedema, excluding chronic inducible urticaria and urticarial vasculitis. Among all patients with chronic urticaria, CSU patients accounts for about 80%. Although the pathogenesis of CSU is still unclear, increasing evidence has shown an autoimmune feature of this chronic disease. Oral antihistamines are the mainstay of treatment for patients with CSU. However, a proportion of patients with CSU remain symptomatic despite treatment with standard- or doubled-dose of antihistamines. In recent years, studies have shown that low-dose recombinant human IL-2 (rhIL-2) treatment has good therapeutic effect in a variety of autoimmune diseases, such as systemic lupus erythematosus, type 1 diabetes, without serious side reactions. Therefore, we propose low-dose rhIL-2 as an add-on treatment for patient with CSU that are recalcitrant to treatment with antihistamines. Here we designed this clinical trial to explore its therapeutic effect as well as therapeutic mechanisms.

Design of Study:

This is a randomized, controlled, single-center clinical trial to assess the short-term efficacy of rhIL-2 treatment for patients with CSU.

Methods:

RhIL-2 injection combined with the current dose of antihistamine (Use one kind or two to three kinds in combination, and use one or two doses of each kind of antihistamine，keeping doses before enrollment) will be applied to CSU patients meeting the inclusion criteria. The end points include clinical response and immunological changes, as well as safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age: between 18- and 75-years old;
2. Patients definitely diagnosed with chronic spontaneous urticaria according to 'Guideline for diagnosis and treatment of urticaria in China (2018) '; or chronic spontaneous urticaria has been diagnosed in the past.
3. Patients taking antihistamines daily ( one kind or two to three kinds in combination, with a standard- or doubled-dose of each kind of antihistamines) for at least one week and remain symptomatic with a UAS7 score of not less than 16;
4. Written informed consent was obtained, and the patient volunteers to participate in the project and complete the project as required.

Exclusion Criteria:

1. Patients with severe diseases of heart, brain, lungs, liver, kidney or blood system; patients experienced organ transplantation;
2. Patients with any acute severe infection such as pyemia and cellulitis, active tuberculosis, or an infection history of human immunodeficiency virus (HIV);
3. Patients have a clear history of allergy to rhIL-2;
4. Patients receiving Interleukin-2 treatment in the last 3 months by subcutaneous or intramuscular injection；
5. Patients with drug abuse, alcohol abuse, or mental disorders that are unable to cooperate or adhere to treatment;
6. Pregnant women, lactating women or women who are willing to conceive within 3 months;
7. Patients receiving glucocorticoid treatment in the last 4 weeks; Patients receiving cyclosporin treatment in the last 90 days；Patients receiving tripterygium wilfordii polyglycoside treatment in the last 6 months；Patients receiving Omalizumab treatment in the last 1 year；Other drugs used previously should be identified whether they are in the washout period one by one, and patients who have taken drugs that may have an impact on the study should be excluded during the washout period or screened again for enrollment after the washout period；
8. Patients who have participated in other clinical trials within 3 months before the screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-06-16 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
The change of Urticaria Activity Score of 7 Days（UAS7）from baseline (Day 0) to Day 14. | from baseline to Day 14
  UAS7 score on Day 14 - UAS7 score on Day 0

SECONDARY OUTCOMES:
The change of UAS7 from baseline (Day 0) to Day 28 and Day 56, respectively. | from baseline to Day 28 and Day 56, respectively
  UAS7 score on Day 28 (or Day 56) - UAS7 score on Day 0
The change of chronic urticaria quality of life questionnaire (CU-Q2oL) score after a 14-, 28- and 56-day treatment, respectively. | from baseline to 14, 28 and 56 days, respectively
  CU-Q2oL score on Day 0 - CU-Q2oL score on Day N
The change of urticaria control test (UCT) after a 14-, 28- and 56-day treatment, respectively. | from baseline to 14, 28 and 56 days, respectively
  UCT score on Day 0 - UCT score on Day N
For patients with angioedema, the change of Angioedema Activity Score of 7days（AAS7）after a 14-, 28- and 56-day treatment, respectively. | from baseline to 14, 28 and 56 days, respectively
  AAS7 on Day 0 - AAS7 on Day N
For patients with angioedema, the change of Angioedema quality of life questionnaire(AE-QoL) after a 28- and 56-day treatment, respectively. | from baseline to 28 and 56 days, respectively
  AE-QoL on Day 0 - AE-QoL on Day N
The change of sera autoantibodies titer after a 14- and 28-day treatment, respectively. | from baseline to 14 and 28 days, respectively
  The autoantibodies including IgG-anti-FcεRⅠand IgG-anti-IgE antibodies titer are detected by Elisa.
The change of accumulative dose of antihistamines in the past 7 days on Day 28 and Day 56, respectively, compared to baseline. | from baseline to 28 and 56 days, respectively
  The accumulative dose of antihistamines in the past 7 days will be calculated on Day 28 and Day 56, respectively, and compared to that of baseline.
Percentage of patients with UAS7 less than 6 on Day 14 and Day 28, respectively. | from baseline to 28 and 56 days, respectively
  The percentage of patients with UAS7 less than 6 were calculated on Day 14 and Day 28, respectively.
The drug adverse reactions throughout the entire study process. | through study completion, an average of 56 days
  The adverse reactions of rhIL-2 including fever, myalgia, nausea, emesis, rash.

CONTACTS AND LOCATIONS:
Overall Officials: Qianjin Lu, MD, PhD, Principal Investigator — The Second Xiangya Hospital, Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China